CLINICAL TRIAL: NCT02370511
Title: The Safety and Feasibility of the SAPIEN XTTM Transcatheter Heart Valve With NovaFlex and Ascendra Delivery Systems and SAPIEN 3 With Commander Delivery System in Patients With Symptomatic Severe Calcific Mitral Valve Disease With Severe Mitral Annular Calcification and Patients With Failing Mitral Surgical Rings or Bioprostheses Who Are Not Candidates for Mitral Valve Surgery.
Brief Title: Mitral Implantation of TRAnscatheter vaLves
Acronym: MITRAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayra Guerrero (Other)
Collaborators: Henry Ford Hospital (Other)
Responsible Party: Sponsor-Investigator, Mayra Guerrero, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-006601
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Results first posted 2021-08-16 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Mitral Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Native mitral valve with severe MAC (Experimental): Patients with symptomatic severe calcific native mitral valve disease with severe mitral annular calcification who have extremely high surgical risk for standard surgical mitral valve replacement, will undergo transcatheter mitral valve replacement.
  Interventions: Device: Transcatheter Mitral Valve Replacement
- Valve-in-Ring (Experimental): Patients with symptomatic failing surgical rings resulting in severe mitral regurgitation or stenosis will undergo transcatheter mitral valve replacement (valve-in-ring).
  Interventions: Device: Transcatheter Mitral Valve Replacement
- Valve-in-Valve (Experimental): Patients with symptomatic failing surgical bioprostheses resulting in severe mitral regurgitation or stenosis will undergo transcatheter mitral valve replacement (Valve-in-valve).
  Interventions: Device: Transcatheter Mitral Valve Replacement

INTERVENTIONS:
Device: Transcatheter Mitral Valve Replacement — Implantation of a balloon expandable Edwards SAPIEN XT or SAPIEN 3 transcatheter heart valve in the mitral position.

SUMMARY:
The purpose of this trial is to establish the safety and feasibility of the Edwards SAPIEN XT™and SAPIEN 3™ device and delivery systems in patients with severe symptomatic calcific mitral valve disease with severe mitral annular calcification who are not candidates for standard mitral valve surgery.

DETAILED DESCRIPTION:
Design:

A prospective pilot study enrolling extremely high surgical risk patients with symptomatic severe calcific mitral valve disease undergoing implantation of an Edwards Sapien XT or SAPIEN 3 valve in the mitral position.

There are three arms in this study evaluating three separate patient populations described below:

* Native Mitral Valve with severe Mitral Annular Calcification (MAC): Patients with symptomatic severe disease of a native mitral valve due to severe mitral annular calcification.
* Valve-in-Ring: Patients with symptomatic failing surgical rings resulting in severe mitral regurgitation or stenosis.
* Valve-in-Valve: Patients with failing bioprosthetic surgical valves with severe regurgitation or stenosis

The delivery approaches include: standard transeptal, modified transeptal approach with a guidewire externalized through a sheath percutaneously placed in the left ventricle, surgical trasnapical and surgical transatrial delivery approach with or without surgical resection of the anterior mitral valve (MV) leaflet (in the native mitral valve arm).

The MITRAL Trial site investigative team (heart team) consists of dedicated representatives from cardiac surgery, interventional cardiology, echocardiology, neurology, study coordination and other multi-disciplinary team members consistent with a transcatheter aortic valve replacement (TAVR) model.

Endpoints

Most endpoints were defined following the Mitral Valve Academic Research Consortium (MVARC) recommendations with minor modifications.73

The primary safety endpoint is: technical success at exit from the cath lab

• Technical success (at exit from the cath lab) is defined as:

* Successful vascular and/or TA access, delivery and retrieval of the transcatheter valve delivery system
* Deployment of a single valve
* Correct position of transcatheter valve in the mitral annulus
* Adequate performance of the prosthetic heart valve (mean mitral valve gradient (MVG) <10 mmHg) without residual mitral regurgitation (MR) grade ≥2 (+)
* No need for additional surgery or re-intervention (includes drainage of pericardial effusion)
* The patient leaves the cath lab alive

The primary performance endpoint is: absence of MR grade 2 (+) or greater or mean MVG ≥10 mmHg at 30 days and 1 year.

Secondary safety endpoints include: Procedural success and all -cause mortality at 30 days and 1 year.

* Procedural Success (30 days) in defined as:

  * Device success at 30 days
  * No device/procedure related severe adverse event (SAE's) including: death, stroke, MI or coronary ischemia requiring PCI or CABG, stage 2 or 3 AKI including dialysis, life threatening bleeding, major vascular or access complications (arterial, venous, or TA - any event requiring additional unplanned surgical or transcatheter intervention), pericardial effusion or tamponade requiring drainage, severe hypotension, heart failure or respiratory failure requiring intravenous pressors or invasive or mechanical treatments such as ultrafiltration or hemodynamic assist devices including intra-aortic balloon pump or left ventricular assist device, or prolonged intubation for ≥48 hrs, or any valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention.
* Device success is defined as:

  * Stroke free survival with original valve in place
  * No need for additional surgery or re-intervention related to the procedure, access or to the replacement valve
  * Proper placement and intended function of the replacement valve, including
  * No migration, fracture, thrombosis, hemolysis or endocarditis
  * No replacement valve stenosis (MV gradient < 10 mmHg)
  * Replacement valve regurgitation < 2 + (including central and paravalvular leak) and without associated hemolysis
  * No increase in AI from baseline (more than 1 grade) and LVOT gradient < 20 mmHg increase from baseline

Additional secondary safety and effectiveness endpoints will be evaluated at two time points: (1) acute, covering events occurring out to 30 days or hospital discharge, whichever is longer; and (2) longer-term, covering events from 31 days to 1 year, and include the following:

Additional Safety Endpoints:

Freedom from

* all stroke and TIA (MVARC)
* myocardial infarction
* major vascular complication (MVARC)
* life-threatening bleeding (MVARC)
* mitral valve reoperation or catheter-based intervention for: valve thrombosis, valve displacement, or other valve placed procedure-related complication
* hemolysis
* endocarditis
* moderate or severe central mitral insufficiency ≥ 2 (+), and/or moderate or severe perivalvular leak causing ≥ 2 (+) mitral insufficiency
* significant mitral stenosis (mean MVG >10 mmHg)
* new permanent pacemaker insertion
* new aortic valve dysfunction (difference greater than 1(+) severity compared with baseline)
* new LVOT gradient ≥ 20 mmHg, or ≥ 20 mmHg increase from baseline LVOT gradient.
* acute kidney injury (MVARC)
* new onset atrial fibrillation
* blood transfusion
* access site infection
* need for iatrogenic ASD closure after index procedure

Additional Effectiveness Endpoints:

1. Rehospitalization at 1 year and Total days alive and out of hospital (from date of index procedure)
2. Clinical improvement per NYHA Class (from baseline) by at least 1 class.
3. Clinical improvement per Quality of Life instruments (>10 points from baseline): (KCCQ 12) (Appendix N)
4. Clinical improvement per 6 Minute Walk Test (> 50 meters from baseline) and 5 meter walk test. (Appendix H)
5. Mean ICU and total index procedure hospital length of stay

Additional Valve Performance Endpoints:

1. Freedom from major mitral paravalvular leak
2. Improvement in hemodynamic function: mean gradient
3. Freedom from structural valve deterioration
4. Total mitral regurgitation

ELIGIBILITY:
Inclusion Criteria in Native Mitral Valve arm

All Candidates must meet the following criteria:

1. Patient has severe calcific native mitral valve stenosis with mitral annular calcification with echocardiographically derived mitral valve area (MVA) of ≤1.5 cm2, or severe mitral regurgitation with severe mitral annular calcification and at least moderate mitral valve stenosis. Qualifying echo must be within 60 days of the date of the procedure.
2. Patient is symptomatic from mitral valve disease, as demonstrated by reported NYHA Functional Class II or greater, or symptoms during stress test.
3. The patient is at least 22 years old.
4. The heart team agrees (and verified in the case review process) that valve implantation will likely benefit the patient.
5. The heart team agrees that medical factors preclude operation, based on a conclusion that the probability of death or serious, irreversible morbidity exceeds the probability of meaningful improvement. Specifically, the STS score is ≥15% or the probability of death or serious, irreversible morbidity is ≥ 50%. The surgeons' consult notes shall specify the medical or anatomic factors leading to that conclusion and include a printout of the calculation of the STS score to additionally identify the risks in the patient (some medical factors and definitions are provided below). At least one of the cardiac surgeon assessors must have physically evaluated the patient. All patients must be approved by the Patient Selection and Procedure Management Steering Committee (at least 2 member votes, one must be a cardiac surgeon).
6. The study patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
7. The study patient agrees to comply with all required post-procedure follow-up visits including annual visits through 5 years and analysis close date visits, which will be conducted as a phone follow-up.

Inclusion Criteria in Valve-in-Ring arm

All Candidates must meet the following criteria:

1. Patient has a failing surgical ring in the mitral position with severe mitral regurgitation or stenosis (echocardiographically derived mitral valve area [MVA] of ≤1.5 cm2. Qualifying echo must be within 60 days of the date of the procedure.
2. Patient is symptomatic from mitral valve disease, as demonstrated by reported NYHA Functional Class II or greater, or symptoms during stress test, or severe hemolytic anemia requiring blood transfusions and no other cause of hemolytic anemia is found after extensive work up.

Inclusion Criteria items #3 to 7 will be the same as in Native MV arm described above

Inclusion Criteria in Valve-in-Valve arm

All Candidates must meet the following criteria:

1. Patient has a failing surgical bioprosthesis in the mitral position with severe mitral regurgitation or stenosis with echocardiographically derived mitral valve area (MVA) of ≤1.5 cm2. Qualifying echo must be within 60 days of the date of the procedure.
2. Patient is symptomatic from mitral valve disease, as demonstrated by reported NYHA Functional Class II or greater, or symptoms during stress test.

Inclusion Criteria items #3 to 7 will be the same as in Native MV arm described above

Exclusion Criteria:

Candidates will be excluded from the study if any of the following conditions are present:

1. Heart Team assessment of operability (the heart team considers the patient is a surgical candidate).
2. Evidence of an acute myocardial infarction ≤ 1 month (30 days) before the intended treatment [defined as: Q wave MI, or non-Q wave MI with total CK elevation of CK-MB ≥ twice normal in the presence of MB elevation and/or troponin level elevation (WHO definition)].
3. Mitral annulus is not calcified (only applies to patients included in Native MV arm).
4. Complex untreated coronary artery disease:

   1. Unprotected left main coronary artery
   2. Syntax score > 32 (in the absence of prior revascularization)
5. Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days of the index procedure (unless part of planned strategy for treatment of concomitant coronary artery disease). Implantation of a permanent pacemaker is not excluded.
6. Any patient with a balloon valvuloplasty (BMV) within 30 days of the procedure (unless BMV is a bridge to procedure after a qualifying ECHO).
7. Patients with planned concomitant surgical or transcatheter ablation for Atrial Fibrillation.
8. Leukopenia (WBC < 3000 cell/mL), acute anemia (Hgb < 9 g/dL), Thrombocytopenia (Plt < 50,000 cell/mL).
9. Hypertrophic obstructive cardiomyopathy (HOCM).
10. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days of screening evaluation.
11. Need for emergency surgery for any reason.
12. Severe ventricular dysfunction with LVEF < 20%.
13. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
14. Active upper GI bleeding within 3 months (90 days) prior to procedure.
15. A known contraindication or hypersensitivity to all anticoagulation regimens, or inability to be anticoagulated for the study procedure.
16. For patients enrolled in the Native MV arm: Native mitral annulus size < 275 mm2 or > 740 mm2 as measured by CT scan.

    For patients in Valve-in-Ring arm: surgical ring with a true mean internal diameter ≤18 mm or ≥ 29 mm or an area < 275 mm2 or > 740 mm2 as measured by CT scan. Caution recommended in:
    * Incomplete bands due to risk of paravalvular leak and risk of LVOT obstruction. Careful measurements by CT and CT-guided procedural planning is recommended.
    * Non-circular rigid or semi-flexible rings (e.g., D-shaped, saddle shaped, etc) due to risk of para-valvular leak and/or out of round or incomplete valve expansion.

    For patients in Valve-in-Valve arm: surgical bioprosthesis with a true internal diameter ≤18 mm or ≥ 29 mm
17. Clinically (by neurologist) or neuroimaging confirmed stroke or transient ischemic attack (TIA) within 6 months (180 days) of the procedure.
18. Estimated life expectancy < 24 months (730 days) due to carcinomas, chronic liver disease, chronic renal disease or chronic end stage pulmonary disease.
19. Expectation that patient will not improve despite treatment of mitral stenosis
20. Active bacterial endocarditis within 6 months (180 days) of procedure.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mayra E. Guerrero, MD, Principal Investigator — Mayo Clinic
Locations (15):
- United States (15):
  - Banner University Medical Center, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - MedStar Washington Medical Center, Washington D.C., District of Columbia
  - Piedmont HealtCare, Atlanta, Georgia
  - Evanston Hospital / North Shore University HealthSystem, Evanston, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guerrero M, Greenbaum A, O'Neill W. First in human percutaneous implantation of a balloon expandable transcatheter heart valve in a severely stenosed native mitral valve. Catheter Cardiovasc Interv. 2014 Jun 1;83(7):E287-91. doi: 10.1002/ccd.25441. Epub 2014 Mar 14. PMID 24532349
- [Background] Sinning JM, Mellert F, Schiller W, Welz A, Nickenig G, Hammerstingl C. Transcatheter mitral valve replacement using a balloon-expandable prosthesis in a patient with calcified native mitral valve stenosis. Eur Heart J. 2013 Sep;34(33):2609. doi: 10.1093/eurheartj/eht254. Epub 2013 Jul 4. No abstract available. PMID 23828829
- [Background] Hasan R, Mahadevan VS, Schneider H, Clarke B. First in human transapical implantation of an inverted transcatheter aortic valve prosthesis to treat native mitral valve stenosis. Circulation. 2013 Aug 6;128(6):e74-6. doi: 10.1161/CIRCULATIONAHA.113.001466. No abstract available. PMID 23918190
- [Background] Fassa AA, Himbert D, Brochet E, Depoix JP, Cheong AP, Alkhoder S, Nataf P, Vahanian A. Transseptal transcatheter mitral valve implantation for severely calcified mitral stenosis. JACC Cardiovasc Interv. 2014 Jun;7(6):696-7. doi: 10.1016/j.jcin.2013.12.204. Epub 2014 May 14. No abstract available. PMID 24835326
- [Background] Ribeiro HB, Doyle D, Urena M, Allende R, Amat-Santos I, Pasian S, Bilodeau S, Mohammadi S, Paradis JM, DeLarochelliere R, Rodes-Cabau J, Dumont E. Transapical mitral implantation of a balloon-expandable valve in native mitral valve stenosis in a patient with previous transcatheter aortic valve replacement. JACC Cardiovasc Interv. 2014 Oct;7(10):e137-9. doi: 10.1016/j.jcin.2014.02.024. Epub 2014 Sep 17. No abstract available. PMID 25240553
- [Background] Ferrari E, Niclauss L, Locca D, Marcucci C. On-pump fibrillating heart mitral valve replacement with the SAPIEN XT transcatheter heart valve. Eur J Cardiothorac Surg. 2014 Apr;45(4):749-51. doi: 10.1093/ejcts/ezt364. Epub 2013 Jul 11. PMID 23847181
- [Background] Himbert D, Bouleti C, Iung B, Nejjari M, Brochet E, Depoix JP, Ghodbane W, Fassa AA, Nataf P, Vahanian A. Transcatheter valve replacement in patients with severe mitral valve disease and annular calcification. J Am Coll Cardiol. 2014 Dec 16;64(23):2557-8. doi: 10.1016/j.jacc.2014.09.047. No abstract available. PMID 25500243
- [Result] Guerrero M, Wang DD, Eleid MF, Pursnani A, Salinger M, Russell HM, Kodali SK, George I, Bapat VN, Dangas GD, Tang GHL, Inglesis I, Meduri CU, Palacios I, Reisman M, Whisenant BK, Jermihov A, Kaptzan T, Lewis BR, Tommaso C, Krause P, Thaden J, Oh JK, Douglas PS, Hahn RT, Leon MB, Rihal CS, Feldman T, O'Neill WW. Prospective Study of TMVR Using Balloon-Expandable Aortic Transcatheter Valves in MAC: MITRAL Trial 1-Year Outcomes. JACC Cardiovasc Interv. 2021 Apr 26;14(8):830-845. doi: 10.1016/j.jcin.2021.01.052. PMID 33888229
- [Result] Guerrero M, Wang DD, Pursnani A, Salinger M, Russell HM, Eleid M, Chakravarty T, Ng MH, Kodali SK, Meduri CU, Pershad A, Satler L, Waksman R, Palacios I, Smalling R, Reisman M, Gegenhuber M, Kaptzan T, Lewis B, Tommaso C, Krause P, Thaden J, Oh J, Douglas PS, Hahn RT, Kar S, Makkar R, Leon MB, Feldman T, Rihal C, O'Neill WW. Prospective Evaluation of TMVR for Failed Surgical Annuloplasty Rings: MITRAL Trial Valve-in-Ring Arm 1-Year Outcomes. JACC Cardiovasc Interv. 2021 Apr 26;14(8):846-858. doi: 10.1016/j.jcin.2021.01.051. PMID 33888230
- [Result] Guerrero M, Pursnani A, Narang A, Salinger M, Wang DD, Eleid M, Kodali SK, George I, Satler L, Waksman R, Meduri CU, Rajagopal V, Inglessis I, Palacios I, Reisman M, Eng MH, Russell HM, Pershad A, Fang K, Kar S, Makkar R, Saucedo J, Pearson P, Bokhary U, Kaptzan T, Lewis B, Tommaso C, Krause P, Thaden J, Oh J, Lang RM, Hahn RT, Leon MB, O'Neill WW, Feldman T, Rihal C. Prospective Evaluation of Transseptal TMVR for Failed Surgical Bioprostheses: MITRAL Trial Valve-in-Valve Arm 1-Year Outcomes. JACC Cardiovasc Interv. 2021 Apr 26;14(8):859-872. doi: 10.1016/j.jcin.2021.02.027. PMID 33888231
- [Result] Guerrero ME, Eleid MF, Wang DD, Pursnani A, Kodali SK, George I, Palacios I, Russell H, Makkar RR, Kar S, Satler LF, Rajagopal V, Dangas G, Tang GHL, McCabe JM, Whisenant BK, Fang K, Balan P, Smalling R, Kaptzan T, Lewis B, Douglas PS, Hahn RT, Thaden J, Oh JK, Leon M, O'Neill W, Rihal C. 5-Year Prospective Evaluation of Mitral Valve-in-Valve, Valve-in-Ring, and Valve-in-MAC Outcomes: MITRAL Trial Final Results. JACC Cardiovasc Interv. 2023 Sep 25;16(18):2211-2227. doi: 10.1016/j.jcin.2023.06.041. PMID 37758379
- [Derived] Sticchi A, Reineke D, Praz F, Windecker S. Transcatheter Mitral Valve Replacement for Mitral Valve-in-Valve, Valve-in-Ring, and Valve-in-MAC Using Balloon-Expandable Transcatheter Heart Valves. JACC Cardiovasc Interv. 2021 Apr 26;14(8):873-878. doi: 10.1016/j.jcin.2021.02.034. No abstract available. PMID 33888232
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Native Mitral Valve With Severe MAC | Valve-in-Ring | Valve-in-Valve
Started | 31 | 30 | 30
Completed | 19 | 19 | 29
Not Completed | 12 | 11 | 1
Not completed — Death | 10 | 7 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Native Mitral Valve With Severe MAC | Valve-in-Ring | Valve-in-Valve | Total
Number analyzed (Participants) | 31 | 30 | 30 | 91
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 74.5 [71.3 to 81.0] | 71.5 [67.0 to 76.8] | 77.5 [70.3 to 82.8] | 75.5 [67.75 to 82.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 11 | 19 | 52
  Male | 9 | 19 | 11 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 30 | 28 | 30 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 4 | 6
  White | 31 | 27 | 25 | 83
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 30 | 91

OUTCOME MEASURES:

1. Primary Outcome: Technical Success at Exit From the Cath Lab.
Description: Number of subject to achieve technical success (at exit from cath lab) is defined as:
  * Successful vascular delivery and retrieval of transcatheter valve delivery system
  * Deployment of single valve
  * Correct position of transcatheter valve
  * Adequate performance of prosthesis (MVA > 1.5 cm2) without residual MR grade ≥2 (+)
  * No need for additional surgery or re-intervention
  * Patient leaves cath lab alive
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Native Mitral Valve With Severe MAC | Valve-in-Ring | Valve-in-Valve
Number analyzed (Participants) | 31 | 30 | 30
Participants | 23 | 20 | 30

2. Primary Outcome: Absence of MR Grade 2 (+) or Greater
Description: Number of subjects to have absence of MR grade 2 (+) or greater assessed with echocardiography. MR severity grading system ranging from Grade 1=mild; Grade 4=severe.
Time Frame: 30 days and 1 year
Population: For MAC arm at 30 days 5 patients died and one withdrew consent and at 1 yr 5 additional patients died, 1 additional withdrew consent and 1 additional did not complete 1 yr follow up. For Valve-in-Ring arm at 30 days 2 patients died and at 1 yr 5 additional patients died, 1 patient lost to follow up and 3 did not complete 1 yr follow up. For Valve-in-Valve arm 1 patient died. Data was not collected or analyzed for these patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Native Mitral Valve With Severe MAC | Valve-in-Ring | Valve-in-Valve
Number analyzed (Participants) | 25 | 28 | 29
Participants
  30 days | 23 | 28 | 29
  1 year: number analyzed (Participants) | 18 | 19 | 29
  1 year | 18 | 19 | 29

3. Primary Outcome: Mitral Valve Gradient (MVG)
Description: MVG assessed by echocardiography measured in mmHg
Time Frame: 30 days and 1 year
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Native Mitral Valve With Severe MAC | Valve-in-Ring | Valve-in-Valve
Number analyzed (Participants) | 25 | 28 | 29
mmHg
  30 days | 6.0 [5.2 to 7.8] | 7.6 [5.9 to 9.1] | 6.0 [4.7 to 7.3]
  1 year: number analyzed (Participants) | 18 | 19 | 29
  1 year | 6.1 [5.6 to 7.1] | 6.0 [4.7 to 7.3] | 6.6 [5.5 to 8.9]

4. Secondary Outcome: Procedural Success
Description: Number of subject to have procedural success as defined as no device/procedure related SAE's including: death, stroke, MI or coronary ischemia requiring PCI or CABG, stage 2 or 3 AKI including dialysis, life threatening bleeding, major vascular or access complications (arterial, venous, or TA - any event requiring additional unplanned surgical or transcatheter intervention), pericardial effusion or tamponade requiring drainage, severe hypotension, heart failure or respiratory failure requiring intravenous pressors or invasive or mechanical treatments such as ultrafiltration or hemodynamic assist devices including intra-aortic balloon pump or left ventricular assist device, or prolonged intubation for ≥48 hrs, or any valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention.
Time Frame: 30 days
Population: For MAC arm 1 withdrew consent data was not collected or analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Native Mitral Valve With Severe MAC | Valve-in-Ring | Valve-in-Valve
Number analyzed (Participants) | 30 | 30 | 30
Participants | 16 | 22 | 28

ADVERSE EVENTS:
Time Frame: Adverse events were collected all subjects from baseline to end of study, approximately one year.
Arm/Group | Native Mitral Valve With Severe MAC | Valve-in-Ring | Valve-in-Valve
All-Cause Mortality (participants affected / at risk) | 10/31 | 7/30 | 1/30
Serious Adverse Events (participants affected / at risk) | 18/31 | 13/30 | 8/30
Other Adverse Events (participants affected / at risk) | 17/31 | 12/30 | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Native Mitral Valve With Severe MAC (N=31) | Valve-in-Ring (N=30) | Valve-in-Valve (N=30)
Stroke (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 5 (5) | 4 (4) | 0 (0)
Vascular complications (Vascular disorders) | 1 (1) | 2 (2) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 1 (1) | 0 (0)
Hemolytic anemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 0 (0)
Valve thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve reintervention after index procedure (Cardiac disorders) | 4 (4) | 3 (4) | 0 (0)
New permanent pacemaker requirement (Cardiac disorders) | 5 (5) | 0 (0) | 1 (1)
New rehospitalization for heart failure (Cardiac disorders) | 11 (15) | 5 (6) | 5 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Native Mitral Valve With Severe MAC (N=31) | Valve-in-Ring (N=30) | Valve-in-Valve (N=30)
Blood transfusion (Blood and lymphatic system disorders) | 17 (17) | 12 (12) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT02370511/Prot_SAP_000.pdf